CLINICAL TRIAL: NCT01294956
Title: A Clinical Evaluation of an Investigational Lubricant Eye Gel (FID 115958D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-043
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye; artificial tears; corneal staining
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 115958D (Experimental): Lubricant Eye Drop
  Interventions: Other: Lubricant Eye Drop
- Refresh Liquigel (Active Comparator): Lubricant Eye Drop
  Interventions: Other: Refresh Liquigel

INTERVENTIONS:
Other: Lubricant Eye Drop — 1 drop in each eye, four times a day for 42 days
  Arms: FID 115958D
Other: Refresh Liquigel — 1 drop in each eye, four times a day for 42 days
  Arms: Refresh Liquigel

SUMMARY:
The purpose of this study is to estimate the change in sodium fluorescein staining, as a sign of dry eye, during six weeks of treatment with FID 115958D or Refresh Liquigel.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye
* NaFl Corneal staining sum score ≥ 3 in either eye
* Current use of a lubricant eye gel or ointment at least once per week (over the previous month)

Exclusion Criteria:

* No contact lenses wear throughout the study period
* Must not have had punctal plugs inserted within 30 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Corneal Staining | Day 42

REFERENCES:
- [Result] Cohen S, Martin A, Sall K. Evaluation of clinical outcomes in patients with dry eye disease using lubricant eye drops containing polyethylene glycol or carboxymethylcellulose. Clin Ophthalmol. 2014;8:157-64. doi: 10.2147/OPTH.S53822. Epub 2013 Dec 31. PMID 24403819